CLINICAL TRIAL: NCT06346301
Title: Imagery Rescripting for Obsessive Compulsive Disorder and Body Dysmorphic Disorder: a Multiple-Baseline Single-Case Experimental Design.
Brief Title: Imagery Rescripting as a Stand-alone Treatment for OCD and BDD.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Judy Luigjes, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL83374.018.23
Record Dates: First submitted 2024-02-12; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Obsessive-Compulsive Disorder; Body Dysmorphic Disorders; Anxiety Disorders
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Body Dysmorphic Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Multiple baseline case series design: Patients wil be randomized to different lengths of baseline period and the effectiveness of the treatment is tested by comparing means and slopes of daily reported schema- or core beliefs and OCD and BDD severity,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imagery Rescripting (Experimental): Baseline consists of a random assigned period of 3-8 weeks with measurements and no intervention.
  Intervention consists of a maximum of 12 sessions of imagery rescripting, provided twice-weekly.
  Post treatment follow up consists of 6 weeks with only measurements and no intervention.
  Interventions: Behavioral: Imagery rescripting

INTERVENTIONS:
Behavioral: Imagery rescripting — In Imagery Rescripting participants imagine a different sequence of events based on missed emotional needs and rescript until needs are fulfilled. Duration of sessions is up to 90 minutes.

SUMMARY:
The goal of this multiple baseline case series study is to test the effect of imagery rescripting (ImRs) in Obsessive Compulsive Disorder (OCD) and Body Dysmorphic Disorder (BDD).

Primary objective :The course of schema or core beliefs and change in OCD and BDD. To investigate the effectiveness of imagery rescripting on factors presumed to underlie the disorder, according to schema theory, and on OCD and BDD symptoms.

Secondary objective: The change in OCD and BDD symptoms (full questionnaire), schemata and modes, core emotions, mood, affect and obtrusiveness of intrusion.

Other objectives are research into the working mechanisms of imagery rescripting by collecting qualitative data from patients and their practitioner in a qualitative interview.

For this study, a multiple-baseline single-case experimental design (SCED) is used testing different outcome variables in 18 OCD patients and 18 BDD patients. After a variable baseline period of 3-8 weeks participants will start twice weekly with imagery rescripting for 12 sessions, followed by a 6 week follow up.

Participants will rate schema- or core beliefs and OCD or BDD severity on a visual analogue scale. In addition participants will rate core emotions, affect and obtrusiveness of the intrusion. Secondary we will asses four times questionnaires about OCD of BDD symptoms, depression and schemas en modes. After treatment participants will be interviewed about their experiences.

DETAILED DESCRIPTION:
In a multiple baseline case series study the effectiveness of Imagery Rescripting (ImRs) as a treatment for Body Dysmorphic Disorder (BDD) and Obsessive Compulsive Disorder (OCD) will be researched. 18 participants with OCD and 18 participants with BDD will be randomized to a waiting list with variable length between 3-8 weeks. After this participants will enter a 1-3 session for preparation followed by 12 sessions with ImRs, given twice-weekly. Follow up assessment will take place 6 weeks after ending treatment. Primary outcome is schema of core beliefs and OCD or BDD symptoms, operationalized by daily measures with visual analogue scales. Also 4 times the investigator measures the OCD or BDD symptoms with the Yale Brown Obsessive Compulsive Scale (Y-BOCS), depression with the Hamilton Depression Rating Scale (HDRS) and 3 times the schema and mode questionnaires with the Young Schema Questionnaire (YSQ) and de Schema Mode Inventory (SMI). The hypothesis is that the primary outcomes will reduce more during the intervention phase compared to the baseline phase and remain stable or even further improve in the follow-up phase. For the secondary outcomes the investigator hypothesized a decrease in depressive symptoms, a decrease in the emotions guilt or shame and first an increase in sadness, fear and angriness followed by an decrease. The largest effect is expected from pre- to post treatment, with a relative stable little change during baseline and follow-up.

Results will be analyzed using visual inspection, repeated measures ANOVA and multilevel analysis, pooling the effects of the individual cases. Finally, participants will be interviewed post treatment about their experiences during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for OCD or BDD, a primary diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Are aged 18 and beyond
* Dutch literacy
* Cut-off Y-BOCS of 20
* No change in medication. Stable dose at least 6 weeks prior to study.

Exclusion Criteria:

* Current (hypo)mania
* Active suicidal plans
* Current psychosis (excluding delusional symptoms related to disorder)
* Alcohol or drugs abuse as diagnosed by Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Electroconvulsive therapy in last 6 months
* Neurological disorder or Intelligence Quotient < 80

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Schema of core beliefs | 15-22 weeks
  Idiosyncratic schema- or core beliefs related to Obsessive Compulsive Disorder (OCD) or Body Dysmorphic Disorder (BDD) are daily rated on a Visual Analogue Scales (VAS). The mean of the scores is calculated, range 0-100. A higher score indicates symptom severity.
Obsessive Compulsive (OCD) and Body Dysmorphic (BDD)symptoms | 15-22 weeks
  OCD and BDD severity is assessed with items based on the Yale Brown Obsessive Compulsive Scale (Y-BOCS(-BDD)) rated on a Visual Analogue Scale. The mean of the scores is calculated, range 0-100. A higher score indicates symptom severity.

SECONDARY OUTCOMES:
Core Emotions, affect strength, obtrusiveness of intrusion. | 4 times: at start, end baseline (up to 8 weeks), after treatment (expected 6-7 weeks after start intervention), at follow up (6 weeks after ending treatment)
  Rated on a Visual Analogue Scale. The mean of the scores is calculated, range 0-100. A higher score indicates symptom severity.
Yale Brown Obsessive Compulsive Scale (Y-BOCS(-BDD)) | 4 times: at start, end baseline (up to 8 weeks), after treatment (expected 6-7 weeks after start intervention), at follow up (6 weeks after ending treatment)
  Y-BOCS(-BDD) assesses severity of OCD or BDD symptoms. The minimum score is 0, the maximum score is 48. A higher score indicates symptom severity.
Hamilton Depression Rating Scale (HDRS) | 4 times: at start, end baseline (up to 8 weeks), after treatment (expected 6-7 weeks after start intervention), at follow up (6 weeks after ending treatment)
  The Hamilton Depression Rating Scale assesses severity of depression. The minimum score is 0, the maximum score is 52. A higher score indicates symptom severity.
Young Schema Questionnaire (YSQ) and Schema Mode Inventory (SMI) | At start, after treatment (expected 6-7 weeks after start intervention), at follow up (6 weeks after ending treatment)
  The Young Schema Questionnaire and the Schema Mode Inventory assesses severity of schemas and modi. The minimum score per scale is 0, the maximum score is 6. A higher score indicates symptom severity..

OTHER OUTCOMES:
Qualitative interview | Post treatment up to 8 months
  With an interview, participants will be interviewed after treatment. A qualitative analysis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Damiaan Denys, Prof., Principal Investigator — Amsterdam UMC; Arnoud Arntz, Prof., Principal Investigator — Amsterdam UMC
Locations (1):
- Department of Psychiatry, AMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to privacy regulations patient data will not be shared unless the European Union (EU) regulations on data protection are guaranteed.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT06346301/Prot_SAP_ICF_000.pdf